CLINICAL TRIAL: NCT05467553
Title: An Open-label, Randomized Study to Compare the Efficacy and Safety of P1101 Plus Tenofovir Alafenamide With or Without Ursodeoxycholic Acid in Patients With Chronic Hepatitis B and Hepatitis D Virus Co-Infection
Brief Title: A Study to Compare P1101 Plus TAF With or Without UDCA in Patients With HBV and HDV Co-Infection
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: PharmaEssentia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202108021MIPD; P1101-HDV (Other: PharmaEssentia Corporation)
Record Dates: First submitted 2022-07-15; First posted 2022-07-20 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-07

CONDITIONS: Hepatitis D
Keywords: Ropeginterferon alpha-2b, Hepatitis D, UDCA, TAF
MeSH Terms: conditions — Hepatitis D | interventions — Ursodeoxycholic Acid; tenofovir alafenamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAF and P1101 combination therapy with UDCA (Experimental): Ursodeoxycholic Acid (UDCA) 15 mg/kg orally (PO) QD plus TAF 25 mg orally (PO) QD for 60 weeks, with P1101 450 µg subcutaneously (SC) Q2W add-on at treatment week 12 for 48 weeks.
  Interventions: Drug: Ursodeoxycholic acid; Drug: Ropeginterferon alfa-2b; Drug: Tenofovir Alafenamide
- TAF and P1101 combination therapy without UDCA (Active Comparator): TAF 25 mg orally (PO) QD for 60 weeks with P1101 450 µg sub-cutaneously (SC) Q2W add-on at treatment week 12 for 48 weeks.
  Interventions: Drug: Ropeginterferon alfa-2b; Drug: Tenofovir Alafenamide

INTERVENTIONS:
Drug: Ursodeoxycholic acid — Ursodeoxycholic Acid 15 mg/kg PO QD for 60 weeks
  Other Names: Uroso Tablets
  Arms: TAF and P1101 combination therapy with UDCA
Drug: Ropeginterferon alfa-2b — P1101 450 µg SC Q2W add-on at treatment week 12 for 48 weeks
  Other Names: BESREMI
Drug: Tenofovir Alafenamide — TAF 25 mg PO QD for 60 weeks
  Other Names: Vemlidy

SUMMARY:
This is an open-label, randomized, multi-center study in patients with chronic HBV and HDV co-infection.

DETAILED DESCRIPTION:
There will be 2 treatment groups in this study, 15 subjects per group as follows:

Group 1: TAF 25 mg orally (PO) QD for 60 weeks with P1101 450 µg subcutaneously (SC) Q2W add-on at treatment week 12 for 48 weeks.

Group 2: Ursodeoxycholic Acid (UDCA)* 15 mg/kg orally (PO) QD plus TAF 25 mg orally (PO) QD for 60 weeks, with P1101 450 µg subcutaneously (SC) Q2W add-on at treatment week 12 for 48 weeks.

Both groups will have a post-treatment follow-up of 24 weeks.

*: Dose of Ursodeoxycholic Acid (UDCA) will be determined by weight at Day 1 (TW0) in 2-4 divided doses.

ELIGIBILITY:
Inclusion Criteria:

1. Positive for HBsAg for at least 6 months, either HBeAg(+) or HBeAg(-), and positive for anti-HDV with detectable HDV RNA and ALT ≥ ULN to ≤ 10X ULN at screening.
2. Interferon treatment naïve.
3. Willing and able to provide written informed consent.
4. Age 20-75 years old; subjects who are over 70 years of age must be in generally good health.
5. Laboratory test results before study entry: WBC ≥ 3,000/mm3; ANC ≥ 1,500/mm3; Platelet ≥ 90,000/mm3; Hemoglobin ≥ 10g/dL; e-GFR ≥ 60mL/min.
6. ECG without clinically significant abnormalities before study entry.
7. Be able to attend all scheduled visits and to comply with all study procedures.
8. Patients with anti-HCV(+) or anti-HIV(+) can be enrolled if:

   1. anti-HCV(+) with undetectable HCV RNA ≥ 3 months.
   2. anti-HIV(+) with undetectable HIV viral load (either with or without Highly Active Anti- Retroviral Therapy, HAART).

Exclusion Criteria:

1. Clinically significant illness or surgery that might interfere with study participation.
2. Clinically significant vital sign abnormalities, uncontrolled hypertension, or fever [body temperature >38 degrees Celsius].
3. History of significant alcohol or drug abuse within 6 months prior to the screening visit (alcohol consumption of more than 14 units of alcohol per week [1 Unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol]) or refusal to abstain from alcohol or illicit drugs throughout the study.
4. Any history or presence of poorly controlled or clinically significant medical conditions that are not suitable to receive interferon-based treatment, at the discretion of the investigator: major psychiatric (including but not limited to those with severe depression, severe bi-polar disorder, schizophrenia, suicidal ideation or history of suicidal attempt), neurological, cardiovascular, pulmonary, hematologic, immunologic, autoimmune diseases, thyroid or other endocrine diseases, metabolic (e.g. diabetes mellitus with HbA1C > 8.0%) or other uncontrolled systemic disease, coagulation disorders or blood dyscrasias.
5. Pregnant subject; female subject who are breast feeding or lactating; female subject or the spouse of male subject, with child-bearing potential who is unwilling or unable to practice adequate contraception, defined as vasectomy in men, tubal ligation in women, or use of condoms and spermicides, or birth control pills, or intrauterine devices throughout the study.
6. History of severe allergic or hypersensitivity reactions, e.g. hypersensitivity to the active substance or to any of the excipients of ropeginterferon alfa 2b, ursodeoxycholic acid, tenofovir disoproxil fumarate and tenofovir alafenamide.
7. Therapy with any systemic anti-viral treatment, anti-neoplastic, or immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) within 1 month (3 months for those with long elimination half-lives) prior to the first dose of study drug.
8. A depot injection or an implant of any drug within 3 months prior to administration of study medication, other than contraception or hyaluronic acid injections in joints for osteoarthritis.
9. Body organ transplant or taking immunosuppressant.
10. Use of an investigational drug within 4 weeks prior to the first dose of the study drug.
11. History of malignancy diagnosed or treated within 5 years prior to screening (except for localized treatment of squamous or non-invasive basal cell skin cancers; cervical carcinoma in situ); cancer survivors not on maintenance therapy within the past 5 years.
12. History of opportunistic infection (e.g., invasive candidiasis or pneumocystis pneumonia).
13. Serious localized infection (e.g., cellulitis, abscess) or systemic and life-threatening infection (e.g., septicemia) within 3 months prior to screening.
14. Clinically significant medical conditions known to interfere absorption, distribution, metabolism or excretion of the study drugs.
15. Decompensated liver disease, which includes but not limited to the following: total bilirubin ≥ 2 mg/dL (except in Gilbert syndrome), direct bilirubin ≥ 2X ULN, albumin level < 3.5 g/dL, INR ≥ 1.5; clinical evidence of ascites, liver decompensation, hepatic encephalopathy, oesophageal varices or cirrhosis as identified by ultrasound or any other examination before study entry.
16. Significant steatohepatitis by ultrasound or other examination at the discretion of investigator.
17. Other form of significant chronic liver diseases, except those mentioned above.
18. Significant or major fundoscopic findings at screening including but not limited to retinal exudates, hemorrhage, detachment, neovascularization, papilloedema, optic atrophy, microaneurysms and macu-lar changes.
19. Patients with complete biliary obstruction, chololithiasis, severe pancreatic disease or peptic ulcer.
20. Patients treated by monotherapy of telbivudine/TDF/TAF/adefovir dipivoxil or any other combination therapy with telbivudine/TDF/TAF/adefovir dipivoxil within 1 month prior to screening.
21. Patient who vaccination with any live attenuated vaccine within 1 month prior to screening.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-24 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
HDV RNA level | Week 60
  Decline in HDV RNA ≥ 2 log10 IU/mL at Week 60
ALT level | Week 60
  ALT normalization (ALT < upper limit of normal) at Week 60

SECONDARY OUTCOMES:
Undetectable HDV RNA | Week 60 and Week 84
  Undetectable HDV RNA (HDV RNA< low limit of quantifica-tion) at Week 60 and Week 84
HBsAg level | Week 60 and Week 84
  Reduction in HBsAg ≥ 1 log10 IU/mL at Week 60 and Week 84
Undetectable HBsAg | Week 60 and Week 84
  HBsAg loss at Week 60 and Week 84
HBsAg and anti-HBs level | Week 60 and Week 84
  HBsAg seroconversion (HBsAg loss plus positive anti-HBs) at Week 60 and Week 84
HDV RNA level | Week 84
  Decline in HDV RNA ≥ 2 log10 IU/mL at Week 84
ALT level | Week 84
  ALT normalization (ALT < upper limit of normal) at Week 84

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Jer Chen, Principal Investigator — National Taiwan University Hospital
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No